CLINICAL TRIAL: NCT04799782
Title: Role of Mirtazapine in Ameliorating Sleep Disordered Breathing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Dr. Abdulghani Sankari, MD PhD, Professor, Clinical Educator, Pulmonary/Critical Care Fellowship Program Director, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 100712M1F(V)
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injuries; Sleep Disordered Breathing
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea Syndromes | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirtazapine (Active Comparator): The drug will be taken for a one week peroid.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): The drug will be taken for a one week peroid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — 15 mg dose before bed-time
  Arms: Mirtazapine
Drug: Placebo — One placebo pill before bed-time
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at the effect of using Mirtazapine to target a specific pathway in the body, that relies on a natural chemical the body produces called 'serotonin', in patients with spinal cord injury (SCI) and non-injured persons during sleep. During this part of the study participants will be asked to take Mirtazapine (15mg per day) and a placebo in a random fashion, each for a one week period (drug period) of time followed by one week without drugs (washout period). The drugs will not be taken all at the same time, but each will be taken separately for one weeks followed by a night study to look at the effect the Mirtazapine/placebo pill has on the way the body responds during sleep.

DETAILED DESCRIPTION:
Randomized placebo controlled cross-over study. Each subject will be studied on two separate occasions: (1) Mirtazapine vs. placebo for one week; the participants will be blinded to whether they are taking Mirtazapine or placebo. After the one week treatment a sleep study will be repeated. Mirtazapine will be given at 15 mg dose before bed-time. (2) Cross over medication for one week will be followed by a second sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with SCI (>6months after spinal cord injury) at the T6 level/above
* Non-injured adults

Exclusion Criteria:

* Pregnant and lactating females
* Heart failure, vascular disease, or stroke
* Advanced chronic obstructive pulmonary disease (COPD), liver disease, and chronic kidney disease
* BMI >38 kg/m2
* Mechanical ventilation dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the primary site at John D. Dingell VA Medical Center.
Pre-assignment Details: Of 150 available, 18 participants were enrolled. Of the 18 enrolled, 15 started the study protocol. Of the 15 that started the study protocol, 10 completed the study and had their results analyzed.
Groups:
- Placebo->Mirtazapine: Participants first received a placebo taken once daily for one week. After a washout period of one week, the participants then received mirtazapine taken once daily (15 mg) for one week.
- Mirtazapine->Placebo: Participants first received mirtazapine taken once daily (15 mg) for one week. After a washout period of one week, the participants then received a placebo taken once daily for one week.
Period: First Intervention
Arm/Group | Placebo->Mirtazapine | Mirtazapine->Placebo
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout
Arm/Group | Placebo->Mirtazapine | Mirtazapine->Placebo
Started | 8 | 7
Completed | 6 | 4
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention
Arm/Group | Placebo->Mirtazapine | Mirtazapine->Placebo
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Mirtazapine (15 mg) or Placebo tablet
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: CO2 Reserve (Delta-PETCO2-AT)
Description: Randomized placebo-controlled cross-over study. Each subject was studied on two separate occasions: (1) Mirtazapine vs. placebo for one week; After the one-week treatment a physiological sleep study was performed to determine the CO2 reserve (Delta-PETCO2-AT) and hypocapnic apneic threshold. (2) Cross over medication for one week was followed by a second physiological sleep study to determine the CO2 reserve (Delta-PETCO2-AT) and hypocapnic apneic threshold.
Time Frame: One Week
Population: Only 10 of the 15 enrolled participants finished both medication arms (placebo, mirtazapine) and were used in the final analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 10 | 10
mmHg | -3.8 (1.2) | -2.0 (1.5)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; Test type: Superiority; p = 0.015, t-test, 2 sided

2. Secondary Outcome: AHI (Apnea/Hypopnea Index)
Description: AHI is an index that measures the severity of sleep apnea and is calculated by dividing the total number of apneas and hypopneas by the number of hours of sleep. Randomized placebo-controlled cross-over study. Each subject was studied on two separate occasions: (1) Mirtazapine vs. placebo for one week; After the one-week treatment a polysomnogram (PSG) study was performed to determine the AHI. (2) Cross over medication for one week was followed by a second PSG to determine the AHI.
Time Frame: One Week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events/Hour
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 10 | 10
Events/Hour | 46.4 (22.5) | 47.8 (20.6)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; Test type: Superiority; p = 0.82, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the one-week interventions during which the participants were taking Mirtazapine or placebo
Description: Of the 15 participants who started the study protocol, 13 received Mirtazapine and 12 received a placebo due to participant withdrawal and physician removal.
Arm/Group | Mirtazapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine (N=13) | Placebo (N=12)
Suicidal Thoughts (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine (N=13) | Placebo (N=12)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* The sample size is small and the majority are males, therefore findings from this study may not be applicable to the general population
* The study required heavy instrumentation which may have affected natural sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT04799782/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT04799782/SAP_001.pdf